CLINICAL TRIAL: NCT01018433
Title: Development of an Intervention for Non-Suicidal Self-Injury in Young Adults
Brief Title: Treatment for Non-Suicidal Self-Injury in Young Adults
Acronym: T-SIB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fordham University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH082824 (NIH); K23MH082824 (NIH); DATR AK-TNAI2 (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Non-suicidal Self-injury
Keywords: self-injury; non-suicidal self-injury; deliberate self-harm; self-mutilation
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T-SIB (Experimental): Treatment for self-injurious behaviors; study intervention
  Interventions: Behavioral: T-SIB
- Treatment as Usual (Other)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: T-SIB — Treatment for self-injurious behaviors; study psychotherapy
  Arms: T-SIB
Other: Treatment as usual — Can include other psychotherapy and pharmacotherapy
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to investigate an intervention specifically for non-suicidal self-injury (NSSI) in young adults. The goal of this 9-session outpatient intervention is to reduce the frequency and severity of NSSI. During Phase I, 12 patients will be treated in an open pilot trial. During Phase II, 60 patients will be treated in a randomized controlled pilot study in order to determine the feasibility and acceptability of the intervention and to investigate change in NSSI frequency and severity over time.

DETAILED DESCRIPTION:
Non-suicidal self-injury (NSSI), deliberate harm to the body without suicidal intent, is highly prevalent in young adults, with 1 in 10 college students engaging in over 100 episodes in their lifetimes. Consequences of NSSI are severe, including physical injury ranging in medical severity, distress from shame associated with the behavior, social isolation, psychological symptoms, and increased risk and lethality of NSSI over time. Despite the prevalence and significant consequences of NSSI, no empirically supported treatments specific to NSSI exist. The purpose of this study is to develop, implement, and evaluate an intervention specifically for NSSI in young adults, the Treatment for Self-Injurious Behaviors (T-SIB). This time-limited intervention will integrate theoretically-based strategies whose utility has been identified through empirical research with the goal of reducing frequency and severity of NSSI. The research plan consists of 2 phases. During Phase 1, 12 patients will be treated in an open pilot trial. During Phase 2, 60 patients will be treated in a randomized controlled pilot study to determine the feasibility and acceptability of T-SIB, investigate change in NSSI frequency and severity between T-SIB and treatment as usual (TAU) through a 3-month follow up period, and evaluate the research design of the randomized controlled pilot study to inform both the utility and design of a larger randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-29
* NSSI within the past month OR history of NSSI and urge to self-injure within the past month

Exclusion Criteria:

* Psychotic symptoms
* Severe suicidal ideation

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
NSSI frequency and severity | Baseline, Mid-Treatment, Post-Treatment, 3-month Follow Up

SECONDARY OUTCOMES:
BDI-II BAI MSI-BPD CSI SPSI-R SCL-90-R URICA | Baseline, Post-Intervention, 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Margaret S Andover, Ph.D., Principal Investigator — Fordham University
Locations (1):
- Fordham University, The Bronx, New York, United States